CLINICAL TRIAL: NCT00905944
Title: Effects of an Exercise Program on the Tendance to Severe Arrhythmias in Patients With Severely Impaired Left Ventricular Function and Cardial Re-synchronisation Therapy
Brief Title: Exercise in Patients With a Biventricular Pacemaker
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Charite University, Berlin, Germany (Other)
Responsible Party: Dr. Fernando Dimeo, Dept. of Sports Medicine, Charité Universitätsmedizin Berlin
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: EA4/063/07
Record Dates: First submitted 2009-05-19; First posted 2009-05-21 (Estimated); Last update posted 2009-12-23 (Estimated); Status verified 2009-12

CONDITIONS: Left Ventricular Failure
Keywords: Left ventricular failure; chronic heart failure; Pacemaker; Resynchronisation therapy; Exercise; Endurance exercise
MeSH Terms: conditions — Heart Failure; Motor Activity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (No Intervention)
- Intervention (Experimental): The patients carry out an exercise program (walking on a treadmill) three times weekly for 12 weeks at a speed corresponding with an intensity of 70% of VO2max.
  Interventions: Other: Endurance exercise

INTERVENTIONS:
Other: Endurance exercise — The patients carry out an exercise program (walking on a treadmill) three times weekly for 12 weeks at a speed corresponding with an intensity of 70% of VO2max.
  Arms: Intervention

SUMMARY:
The investigators will evaluate the effects of an exercise program (walking on a treadmill) on the physical performance, the cardiorespiratory function, the proclivity to heart arrhythmias and the quality of life of patients with severely impaired left ventricular function and a bi-ventricular resynchronization pacemaker.

ELIGIBILITY:
Inclusion Criteria:

* Left ventricular failure
* Resynchronization therapy with a biventricular pacemaker
* Ability to understand written German

Exclusion Criteria:

* Age over 75 years
* Severe cardiac arrhythmia
* All conditions which can be aggravated by an exercise program

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-12; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Maximal oxygen uptake (VO2max) | At recruitment and after 12 weeks

SECONDARY OUTCOMES:
Body mass index (BMI) | At recruitment and after 12 weeks
Brain natriuretic peptide (BNP) | At recruitment and after 12 weeks
Body composition | At recruitment and after 12 weeks
Mood | At recruitment and after 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Fernando Dimeo, MD, Principal Investigator — Charite University, Berlin, Germany
Locations (1):
- Section Sports Medicine, Charité Universitätsmedizin Berlin, Hindenburgdamm 30, Berlin, State of Berlin, Germany